CLINICAL TRIAL: NCT03835559
Title: Randomized Controlled Trial Comparing the Clinical Outcomes After Cyanoacrylate Closure and Surgical Stripping for Incompetent Saphenous Veins
Brief Title: Cyanoacrylate Closure Versus Surgical Stripping for Incompetent Saphenous Veins
Acronym: CASS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyung Hee University Hospital at Gangdong (Other)
Responsible Party: Principal Investigator, Jin Hyun Joh, Associate professor, Kyung Hee University Hospital at Gangdong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-03-030-001
Record Dates: First submitted 2019-02-01; First posted 2019-02-08 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Occlusions Vein; Chronic Venous Insufficiency
Keywords: varicose vein; stripping; endovenous; ablation; Occlusion; quality of life
MeSH Terms: conditions — Varicose Veins; Bites and Stings

STUDY DESIGN:
Intervention Model Description: Multicenter, prospective randomized controlled trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cyanoacrylate closure (Active Comparator): After successful access of target vein and insertion of guidewire under any type of anesthesia, the procedure of cyanoacrylate closure for treatment of incompetent Saphenous Veins is performed. A 5 French introducer and catheter is advanced and positioned 5.0 cm caudal to the junction with proximal saphenous vein compression by the ultrasound probe, two injections of approximately 0.10 mL glue are given 1 cm apart, followed by a 3min period of compression, and then repeat injections and 30sec ultrasound probe and hand compression sequences until the entire length of the target vein is treated. The catheter is removed.
  Interventions: Procedure: Cyanoacrylate closure; Procedure: Surgical stripping
- Surgical stripping (Active Comparator): For treatment of incompetent Saphenous Veins, surgical stripping is performed with a proper incision in the groin, with division and ligation of the saphenous vein and division of all tributaries under all types of anesthesia (general, spinal, regional block, or local anesthesia). The saphenous vein is then removed using a stripper. Compression stocking is apply.
  Interventions: Procedure: Cyanoacrylate closure; Procedure: Surgical stripping

INTERVENTIONS:
Procedure: Cyanoacrylate closure — After successful access of target vein and insertion of guidewire under any type of anesthesia, the procedure of cyanoacrylate closure is performed. A 5 French introducer and catheter is advanced and positioned 5.0 cm caudal to the junction with proximal saphenous vein compression by the ultrasound probe, two injections of approximately 0.10 mL glue are given 1 cm apart, followed by a 3min period of compression, and then repeat injections and 30sec ultrasound probe and hand compression sequences until the entire length of the target vein is treated. The catheter is removed.
  Other Names: Cyanoacrylate closure for incompetent Saphenous vein
Procedure: Surgical stripping — All types of anesthesia (general, spinal, regional block, or local anesthesia) can be used. The surgical stripping is performed with a proper incision in the groin, with division and ligation of the saphenous vein and division of all tributaries. The saphenous vein is then removed using a stripper.
  Other Names: Surgical stripping for incompetent Saphenous vein

SUMMARY:
The purpose of this study is to evaluate the non-inferior, clinical outcomes after cyanoacrylate closure comparing the surgical stripping for incompetent saphenous veins.

DETAILED DESCRIPTION:
Varicose veins are highly prevalent. In western countries, an estimated 23% of adults have varicose veins, and 6% have more advanced chronic venous disease, including skin changes and healed or active venous ulcers. There are several modalities to treat varicose veins. Open surgical treatment with ligation and stripping of the saphenous vein, combined with excision of large varicosities, has been the standard of care for many years. Endovenous thermal ablation by radiofrequency ablation (RFA) or endovenous laser ablation (EVLA) has been shown to be a safe and effective alternatives with high long-term target vein closure rates. Although both techniques have gained broad acceptance in many countries, one major disadvantage of these techniques is the requirement for use of tumescent anesthesia to avoid the thermal injury of the surrounding structures. Cyanoacrylate closure for varicose veins has recently been introduced for treatment of the incompetent saphenous vein.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years of age at the time of enrollment
* Reflux in great saphenous vein greater than 0.5 seconds after distal compression and release or Valsalva's maneuver in the standing or reverse Trendelenburg position
* Diameter of saphenous vein between 2mm to 20mm (with standing position)
* One or more of the following symptoms related to the incompetent saphenous vein: aching, throbbing, heaviness, fatigue, pruritus, night cramps, restlessness, generalized pain or discomfort, swelling
* Clinical, Etiologic, Anatomic, and Pathophysiologic classification of C2 through C5

Exclusion Criteria:

* Previous treatment in targeted vein segment
* Tortuous vein in which the delivery catheter cannot be inserted
* Aneurysm of target vein segment >20 mm
* Daily use of narcotic or nonsteroidal anti-inflammatory pain medications to control pain associated with greater saphenous vein reflux
* Known hypercoagulable disorder
* Active malignancy
* Regular use of systemic anticoagulation
* Current use of systemic anticoagulant
* Previous deep vein thrombosis/pulmonary embolism or active acute superficial thrombophlebitis
* Unable to comply with the schedule and protocol evaluations
* Unable to ambulate
* Currently pregnant or breast feeding
* Known sensitivity to cyanoacrylate adhesives
* Symptomatic peripheral arterial disease with ankle-brachial index <0.9
* Participation in another clinical study that has not reached primary endpoint within 30 days prior to enrollment
* Any condition which in the opinion of the investigator could compromise subject safety or adherence to the protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2019-04-10 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Closure rate of the target vein/ Absence of refluxing vein | 3 months
  The primary endpoint of the study is to evaluate the complete closure of the target vein where complete closure is defined as Doppler ultrasound showing vein closure along entire treated vein segment with no discrete segments of patency exceeding 5cm after cyanoacrylate closure and absence of refluxing vein or residual vein after surgical stripping as read by a qualified site technologist or investigator.

SECONDARY OUTCOMES:
Perioperative pain with visual analog scale | 3 days
  The subject will be asked to rate pain on a 0-10 numeric rating scale. (minimum-0 (best), maximum-10 (worst))
Ecchymosis | 3 days
  The investigator will score the subjects ipsilateral leg of the occurrence of ecchymosis along treated segment, rated on a 0- to 5-point graded scale (0, none; 1, involving <25% of the treatment area; 2, 25%-50%; 3, 50%-75%; 4, 75%-100%; 5, extension above or below the treatment segment)
Venous Clinical Severity Score | 1, 3, 6, 12 and 24 months after treatment
  Severity score on a 0-30 numeric rating scale ((minimum-0 (best), maximum-30 (worst))
Acceptability of Quality of life score | 1, 3, 6, 12 and 24 months after treatment
  The quality of life scores are measured by the Aberdeen Varicose Vein Questionnaire (AVVQ) and EuroQOL five dimensions questionnaire (EQ-5D).
  The AVVQs are scored using a questionnaire. The total score for the 13 questions ranges from 0 to 100 points, with 0 points indicating the best possible quality of life. The EuroQOL is an instrument which evaluates the generic quality of life. The EuroQOL descriptive system is a preference-based measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Respondents can report their perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status).
Satisfaction of the patients: satisfaction rate | 1, 3, 6, 12 and 24 months after treatment
  The subject will be asked to the satisfaction rate by five response categories (strongly agree, agree, uncertain, disagree, strongly disagree) after asking as following: I'm very satisfied with the medical care I receive.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Hyun Joh, MD, PhD, Principal Investigator — Kyung Hee University Hospital at Gangdong, Seoul, Korea
Locations (2):
- South Korea (2):
  - In-Mok Jung, Seoul, Non US/Canada
  - Jin Hyun Joh, Seoul, Non US/Canada

IPD SHARING:
Plan to Share IPD: Undecided
Study protocol

REFERENCES:
- [Result] Kaplan RM, Criqui MH, Denenberg JO, Bergan J, Fronek A. Quality of life in patients with chronic venous disease: San Diego population study. J Vasc Surg. 2003 May;37(5):1047-53. doi: 10.1067/mva.2003.168. PMID 12756353
- [Result] van den Bos R, Arends L, Kockaert M, Neumann M, Nijsten T. Endovenous therapies of lower extremity varicosities: a meta-analysis. J Vasc Surg. 2009 Jan;49(1):230-9. doi: 10.1016/j.jvs.2008.06.030. Epub 2008 Aug 9. PMID 18692348
- [Result] Morrison N, Gibson K, McEnroe S, Goldman M, King T, Weiss R, Cher D, Jones A. Randomized trial comparing cyanoacrylate embolization and radiofrequency ablation for incompetent great saphenous veins (VeClose). J Vasc Surg. 2015 Apr;61(4):985-94. doi: 10.1016/j.jvs.2014.11.071. Epub 2015 Jan 31. PMID 25650040
- [Result] Kolluri R, Gibson K, Cher D, Madsen M, Weiss R, Morrison N. Roll-in phase analysis of clinical study of cyanoacrylate closure for incompetent great saphenous veins. J Vasc Surg Venous Lymphat Disord. 2016 Oct;4(4):407-15. doi: 10.1016/j.jvsv.2016.06.017. Epub 2016 Aug 8. PMID 27638993
- [Result] Chan YC, Law Y, Cheung GC, Ting AC, Cheng SW. Cyanoacrylate glue used to treat great saphenous reflux: Measures of outcome. Phlebology. 2017 Mar;32(2):99-106. doi: 10.1177/0268355516638200. Epub 2016 Jul 9. PMID 27052039